CLINICAL TRIAL: NCT00922181
Title: Single-probe Microwave Ablation of Metastatic Liver Cancer is Highly Variable and Irreproducible
Brief Title: Single-probe Microwave Ablation (MWA) of Metastatic Liver Cancer
Acronym: LiverMWA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: University Hospital Gasthuisberg Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kulasMWA1
Record Dates: First submitted 2009-06-01; First posted 2009-06-17 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Liver Neoplasms
Keywords: malignancy; liver; microwave; surgery
MeSH Terms: conditions — Liver Neoplasms; Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MWA (Experimental): Patients undergoing MWA for hepatic metastases smaller than 3 cm, without underlying liver disease
  Interventions: Device: Microwave ablation
- RFA (Active Comparator): Patients undergoing RFA for hepatic metastases smaller than 3 cm, without underlying liver disease
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Microwave ablation — Liver tumors are destructed/ablated using single-probe microwave energy device
  Other Names: MW ablation antenna (VT2237) and a 915 MHz Valleylab MW generator (VTSYS3; Covidien, Europe NV)
  Arms: MWA
Device: Radiofrequency ablation — Liver tumors are destructed/ablated using radiofrequency energy device
  Arms: RFA

SUMMARY:
Microwave ablation (MWA) is the most recent development in the field of local ablative therapies. The aim of this study was to evaluate the variability and reproducibility of single-probe MWA versus radiofrequency ablation (RFA) of metastatic liver tumours smaller than 3 cm in patients without underlying liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable metastatic liver cancer
* No invasion of major biliary structures
* No invasion of major vascular structures
* ASA score < 4
* WHO score 0-1
* Pre-operative chemotherapy is allowed

Exclusion Criteria:

* Resectable liver metastases
* Life expectancy less than 3 months
* Patients with cardiac pacemaker, cerebral aneurysm clips, implanted electronic instruments or other metal materials
* Coagulopathy with platelet count less than 50000
* Active infectious disease
* Age below 18 years
* Pregnancy of breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Variability of ablation diameters | within the first 7 days and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Hompes R, Fieuws S, Aerts R, Thijs M, Penninckx F, Topal B. Results of single-probe microwave ablation of metastatic liver cancer. Eur J Surg Oncol. 2010 Aug;36(8):725-30. doi: 10.1016/j.ejso.2010.05.013. Epub 2010 Jun 3. PMID 20605397